CLINICAL TRIAL: NCT00652938
Title: Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' HPV Vaccine (580299) Co-administrated With a Commercially Available Vaccine in Healthy Female Adolescents
Brief Title: Evaluation of Immunogenicity and Safety of Human Papillomavirus (HPV) Vaccine Co-administered With Another Vaccine in Healthy Female Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111507
Record Dates: First submitted 2008-03-27; First posted 2008-04-04 (Estimated); Results first posted 2010-08-31 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2017-04

CONDITIONS: Infections, Papillomavirus
Keywords: Co-administration; HPV vaccine; Cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Papillomavirus Vaccines; Engerix-B

ARMS (3):
- Cervarix & Engerix Group (Active Comparator): Subjects received 3 doses of Cervarix™ (Human Papillomavirus [HPV] vaccine) co-administered with Engerix™ (Hepatitis B [HBV] vaccine) according to a 0, 1, 6-month schedule.
  Interventions: Biological: HPV Vaccine (GSK580299) Cervarix TM; Biological: Engerix B
- Cervarix Group (Experimental): Subjects received 3 doses of Cervarix™ (Human Papillomavirus [HPV] vaccine) according to a 0, 1, 6-month schedule.
  Interventions: Biological: HPV Vaccine (GSK580299) Cervarix TM
- Engerix Group (Active Comparator): Subjects received 3 doses of Engerix™ (Hepatitis B [HBV] vaccine) according to a 0, 1, 6-month schedule.
  Interventions: Biological: Engerix B

INTERVENTIONS:
Biological: HPV Vaccine (GSK580299) Cervarix TM — IM administration
  Arms: Cervarix & Engerix Group; Cervarix Group
Biological: Engerix B — IM administration
  Arms: Cervarix & Engerix Group; Engerix Group

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the necessary cause of cervical cancer. Vaccination of pre-teens and adolescents, ideally before sexual debut and thus before exposure to oncogenic HPV, is a rational strategy for prevention of cervical cancer. Thus, HPV vaccination could complement the existing pre-adolescent/adolescent vaccination programs. This Phase IIIb study is designed to evaluate the immunogenicity and safety of co-administering a commercially available vaccine with GSK Biologicals' HPV-16/18 L1 VLP AS04 (Cervarix TM) vaccine as compared to the administration of either vaccine alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parents/legally acceptable representatives (LARs) can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits) should be enrolled in the study.
* A female between, and including, 9 and 15 years of age (has not attained her 16th birthday) at the time of the first vaccination.
* Written informed consent obtained from the subject's parent/LAR prior to the enrolment. In addition, written informed assent must be obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects must not be pregnant. Absence of pregnancy should be verified with a urine pregnancy test.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for at least 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for two months after completion of the vaccination series. Subjects who reach menarche (begin menstruating) during the study, and therefore become of childbearing potential, must agree to follow the same precautions.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period (up to Month 12).
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after each dose of vaccine. Administration of routine vaccines such as meningococcal, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccines up to 8 days before the first dose of study vaccine is allowed.
* Concurrently participating in another clinical study, at any time during the study period (up to the Month 12 telephone contact), in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* A subject planning to become pregnant, likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive precautions during the study period and up to two months after the last vaccine dose.
* Pregnant or breastfeeding women.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* Previous administration of components of the investigational vaccine.
* Previous vaccination against hepatitis B or planned administration of any hepatitis B vaccine other than that foreseen by the study protocol during the study period.
* History of hepatitis B infection.
* Known exposure to hepatitis B within the previous 6 weeks.
* Known acute or chronic, clinically significant neurologic, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* Cancer or autoimmune disease under treatment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 9 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 744 (Actual)
Dates: Start 2008-04-09; Primary Completion 2009-08-28 (Actual); Study Completion 2010-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Netherlands (2):
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
- Sweden (5):
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Luleå
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Norrköping
  - GSK Investigational Site, Skene

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Schmeink C et al. Co-administration of AS04-adjuvanted human papillomavirus-16/18 vaccine with hepatitis B vaccine in healthy female subjects aged 9-15 years. Abstract presented at the 28th Annual Meeting of European Society for Paediatric Infectious Diseases (ESPID). Nice, France, 4-8 May 2010.
- [Background] Schmeink CE, Bekkers RL, Josefsson A, Richardus JH, Berndtsson Blom K, David MP, Dobbelaere K, Descamps D. Co-administration of human papillomavirus-16/18 AS04-adjuvanted vaccine with hepatitis B vaccine: randomized study in healthy girls. Vaccine. 2011 Nov 15;29(49):9276-83. doi: 10.1016/j.vaccine.2011.08.037. Epub 2011 Aug 19. PMID 21856349
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 111507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While the total numbers of subjects enrolled in the study was 744, the total number of subjects that entered the study was 741. The remaining 3 subjects received a subject number but no vaccine dose and were therefore excluded from the analysis and group assignment.
Groups:
- Cervarix&Engerix Group: Subjects received 3 doses of Cervarix™ (Human Papillomavirus [HPV] vaccine) co-administered with Engerix™ (Hepatitis B [HBV] vaccine) according to a 0, 1, 6-month schedule.
Period: Overall Study
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Started | 247 | 247 | 247
Completed | 246 | 240 | 242
Not Completed | 1 | 7 | 5
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 6 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — fear of blood sampling | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group | Total
Number analyzed (Participants) | 247 | 247 | 247 | 741
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (2.17) | 11.3 (2.14) | 11.4 (2.17) | 11.4 (2.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 247 | 247 | 741
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-Hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Above the Cut-off Value for Seroprotection
Description: Only groups which had received the HBV vaccine were included in the analysis.
  Subjects included were seronegative for anti-HBs (antibody titer < 3.3 milli International Units per milliliter (mIU/mL)) prior to vaccination.
  Anti-HBs antibody cut-off value for seroprotection assessed included 10 mIU/mL.
Time Frame: Month 7
Population: The analysis was performed on the According-to-Protocol (ATP) Cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 194 | 0 | 181
Participants | 190 |  | 181

2. Primary Outcome: Number of Subjects With Anti-human Papillomavirus 16 and 18 (Anti-HPV-16 and Anti-HPV-18) Antibody Concentrations Above the Cut-off Value for Seroconversion
Description: Only groups which had received the HPV vaccine were included in the analysis.
  Anti-HPV-16 antibody cut-off value assessed included 8 Enzyme-linked Immunosorbent Assay (ELISA) units per milliliter (EL.U/mL) and anti-HPV-18 antibody cut-off value assessed included 7 EL.U/mL.
  Subjects included were seronegative for anti-HPV-16 (antibody titer < 8 EL.U/mL) and anti-HPV-18 (antibody titer < 7 EL.U/mL) prior to vaccination.
Time Frame: Month 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 207 | 202 | 0
Participants
  Anti-HPV-16: number analyzed (Participants) | 207 | 200 | 0
  Anti-HPV-16 | 205 | 200 |
  Anti-HPV-18: number analyzed (Participants) | 200 | 202 | 0
  Anti-HPV-18 | 199 | 202 |

3. Primary Outcome: Anti-HPV-16/18 Antibody Titres
Description: Antibody titers for Anti-HPV-16 and Anti-HPV-18 are expressed as Geometric Mean Titers (GMTs).
  Only groups which had received the HPV vaccine were included in the analysis.
  Subjects included were seronegative for anti-HPV-16 (antibody titer < 8 EL.U/mL) and anti-HPV-18 (antibody titer < 7 EL.U/mL) prior to vaccination.
Time Frame: Month 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 207 | 202 | 0
EL.U/mL
  Anti-HPV-16: number analyzed (Participants) | 207 | 200 | 0
  Anti-HPV-16 | 19819.8 [16856.9 to 23303.6] | 21712.6 [19460.2 to 24225.6] |
  Anti-HPV-18: number analyzed (Participants) | 200 | 202 | 0
  Anti-HPV-18 | 8835.1 [7636.3 to 10222.1] | 8838.6 [7948.5 to 9828.4] |

4. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations Above the Cut-off Value for Seroconversion
Description: Only groups which had received the HBV vaccine were included in the analysis.
  Subjects included were seronegative for anti-HBs (antibody titer < 3.3 mIU/mL) prior to vaccination.
  Anti-HBs antibody cut-off value for seroconversion assessed included 3.3 mIU/mL.
Time Frame: Month 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 194 | 0 | 181
Participants | 192 |  | 181

5. Secondary Outcome: Anti-HBs Antibody Titres
Description: Antibody titers for anti-HBs are given as Geometric Mean Titers (GMTs) in mIU/mL.
  Only groups which had received the HBV vaccine were included in the analysis.
  Subjects included were seronegative for anti-HBs (antibody titer < 3.3 mIU/mL) prior to vaccination.
Time Frame: Month 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 194 | 0 | 181
mIU/mL | 1280.9 [973.3 to 1685.7] |  | 3107.7 [2473.1 to 3905.1]

6. Secondary Outcome: Number of Subjects With Anti-HPV-16 and Anti-HPV-18 Antibody Concentrations Above the Cut-off Value for Seroconversion
Description: as for outcome 2
Time Frame: Month 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 207 | 201 | 0
Participants
  Anti-HPV-16: number analyzed (Participants) | 207 | 199 | 0
  Anti-HPV-16 | 207 | 199 |
  Anti-HPV-18: number analyzed (Participants) | 200 | 201 | 0
  Anti-HPV-18 | 200 | 201 |

7. Secondary Outcome: Anti-HPV-16/18 Antibody Titres
Description: as for outcome 3
Time Frame: Month 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 207 | 201 | 0
EL.U/mL
  Anti-HPV-16: number analyzed (Participants) | 207 | 199 | 0
  Anti-HPV-16 | 4894.7 [4472.5 to 5356.7] | 5069.2 [4581.2 to 5609.1] |
  Anti-HPV-18: number analyzed (Participants) | 200 | 201 | 0
  Anti-HPV-18 | 4790.4 [4338.9 to 5288.8] | 4663.8 [4228.2 to 5144.3] |

8. Secondary Outcome: Number of Subjects With Anti-Hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Above the Cut-off Value for Seroconversion
Description: as for outcome 4
Time Frame: Month 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 194 | 0 | 178
Participants | 165 |  | 168

9. Secondary Outcome: Number of Subjects With Anti-Hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Above the Cut-off Value for Seroprotection
Description: Only groups which had received the HBV vaccine were included in the analysis.
  Subjects included were seronegative for anti-HBs (antibody titer < 3.3 milli International Units per milliliter (mIU/mL)) prior to vaccination vaccination.
  Anti-HBs antibody cut-off value for seroprotection assessed included 10 mIU/mL.
Time Frame: Month 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 194 | 0 | 178
Participants | 128 |  | 142

10. Secondary Outcome: Anti-HBs Antibody Titers
Description: Anti-HBs antibody titers are given as GMTs in mIU/mL.
  Only groups which had received the HBV vaccine were included in the analysis.
  Subjects included were seronegative for anti-HBs (antibody titer < 3.3 mIU/mL) prior to vaccination.
Time Frame: Month 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 194 | 0 | 178
mIU/mL | 13.6 [11.4 to 16.2] |  | 26.9 [22.1 to 32.8]

11. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms
Description: Solicited local symptoms included injection site pain, redness and swelling.
  Any solicited local symptom is occurence of a symptom regardless of its intensity.
Time Frame: During the 7-day period (Days 0 - 6) following vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 247 | 245 | 246
Participants
  Pain | 244 | 238 | 182
  Redness | 122 | 127 | 63
  Swelling | 120 | 111 | 47

12. Secondary Outcome: Number of Subjects Reporting Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms include injection site pain, redness and swelling.
  Grade 3 pain is pain that prevented normal everyday activities. Grade 3 redness is redness that was > 50 mm. Grade 3 swelling is swelling that was > 50 mm.
Time Frame: During the 7-day period (Days 0-6) following vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 247 | 245 | 246
Participants
  Pain | 54 | 35 | 4
  Redness | 12 | 5 | 1
  Swelling | 17 | 13 | 1

13. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptoms
Description: Solicited general symptoms included arthralgia, fatigue, gastrointestinal, headache, myalgia, rash, temperature in degrees celsius (axillary) and urticaria.
  Any solicited general symptom is the occurence of the symptom regardless of its intensity or relationship to study vaccination.
Time Frame: During the 7-day (Days 0-6) period following vaccination.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 247 | 245 | 246
Participants
  Arthralgia | 31 | 23 | 26
  Fatigue | 130 | 107 | 104
  Gastrointestinal | 65 | 67 | 70
  Headache | 136 | 131 | 129
  Myalgia | 55 | 55 | 53
  Rash | 10 | 14 | 11
  Temperature | 32 | 23 | 36
  Urticaria | 5 | 5 | 6

14. Secondary Outcome: Number of Subjects Reporting Grade 3 Solicited General Symptoms
Description: Solicited general symptoms included arthralgia, fatigue, gastrointestinal, headache, myalgia, rash, temperature in degrees celsius (axillary) and urticaria.
  Grade 3 arthralgia, fatigue, gastrointestinal, headache, myalgia and rash were symptoms that prevented normal activity.
  Grade 3 temperature was temperature > 39 degrees Celsius. Grade 3 urticaria was urticaria distributed on at least 4 body areas.
Time Frame: During the 7-day (Days 0-6) period following vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 247 | 245 | 246
Participants
  Arthralgia | 1 | 0 | 0
  Fatigue | 8 | 8 | 9
  Gastrointestinal | 4 | 6 | 8
  Headache | 13 | 11 | 4
  Myalgia | 2 | 2 | 1
  Rash | 0 | 1 | 0
  Temperature | 3 | 2 | 3
  Urticaria | 0 | 0 | 1

15. Secondary Outcome: Number of Subjects Reporting Related Solicited General Symptoms
Description: Solicited general symptoms included arthralgia, fatigue, gastrointestinal, headache, myalgia, rash, temperature in degrees celsius (axillary) and urticaria.
  Related solicited general symptoms were those symptoms assessed by the investigators as related to the study vaccination.
Time Frame: During the 7-day period (Days 0 - 6) following vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 247 | 245 | 246
Participants
  Arthralgia | 18 | 16 | 12
  Fatigue | 89 | 70 | 51
  Gastrointestinal | 35 | 40 | 25
  Headache | 77 | 71 | 57
  Myalgia | 40 | 40 | 20
  Rash | 8 | 8 | 4
  Temperature | 13 | 10 | 6
  Urticaria | 4 | 4 | 2

16. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Causally Related to Vaccination Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
  Grade 3 AE was an AE that prevented normal activities. Related AE was an AE that was assessed by the investigator as related to the study vaccination.
Time Frame: During the 30-day period (Days 0 - 29) following any vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 247 | 247 | 247
Participants
  Any AEs | 130 | 99 | 99
  Grade 3 AEs | 19 | 19 | 16
  Related AEs | 43 | 19 | 25

17. Secondary Outcome: Number of Subjects Reporting Any and Causally Related to Vaccination Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
  Related SAEs were SAEs assessed by the investigators as related to the vaccination.
  * Grade 3 SAEs were not assessed.
Time Frame: Throughout the active phase of the study (up to Month 7).
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 247 | 247 | 247
Participants
  Any | 2 | 1 | 0
  Related | 0 | 0 | 0

18. Secondary Outcome: Number of Subjects Reporting Any and Causally Related to Vaccination SAEs
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
  * Grade 3 SAEs were not assessed.
Time Frame: Throughout the safety follow-up (month 7 up to Month 12).
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 247 | 247 | 247
Participants
  Any | 1 | 1 | 1
  Related | 0 | 0 | 0

19. Secondary Outcome: Number of Subjects Reporting Medically Significant Conditions
Description: Medically significant conditions (i.e., AEs prompting emergency room or physician visits that are not (1) related to common diseases or (2) routine visits for physical examination or vaccination, or SAEs that are not related to common diseases).
Time Frame: Throughout the active phase of the study (up to Month 7)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 247 | 247 | 247
Participants | 31 | 28 | 22

20. Secondary Outcome: Number of Subjects Reporting Medically Significant Conditions
Description: as for outcome 19
Time Frame: Throughout the safety follow-up (month 7 up to Month 12)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 247 | 247 | 247
Participants | 0 | 2 | 2

ADVERSE EVENTS:
Arm/Group | Cervarix&Engerix Group | Cervarix Group | Engerix Group
Serious Adverse Events (participants affected / at risk) | 3/247 | 2/247 | 1/247
Other Adverse Events (participants affected / at risk) | 246/247 | 239/247 | 222/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix&Engerix Group (N=247) | Cervarix Group (N=247) | Engerix Group (N=247)
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix&Engerix Group (N=247) | Cervarix Group (N=247) | Engerix Group (N=247)
Pain (General disorders) | 244 | 238 | 182
Redness (General disorders) | 122 | 127 | 63
Swelling (General disorders) | 120 | 111 | 47
Arthralgia (General disorders) | 31 | 23 | 26
Fatigue (General disorders) | 130 | 107 | 104
Gastrointestinal (General disorders) | 65 | 67 | 70
Headache (General disorders) | 136 | 131 | 129
Myalgia (General disorders) | 55 | 55 | 53
Rash (General disorders) | 10 | 14 | 11
Temperature (General disorders) | 32 | 23 | 36
Nasopharyngitis (General disorders) | 29 | 27 | 26
Headache (General disorders) | 17 | 19 | 9
Oropharyngeal pain (General disorders) | 13 | 13 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.